CLINICAL TRIAL: NCT06500481
Title: A Phase III Randomized Clinical Trial of Proton Craniospinal Irradiation Versus Involved-Field Radiotherapy for Patients With Breast Cancer or Non-Small Cell Lung Cancer Leptomeningeal Metastasis (Radiate-LM)
Brief Title: Testing Proton Craniospinal Radiation Therapy Versus the Usual Radiation Therapy for Leptomeningeal Metastasis, RADIATE-LM Trial
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NRG-BN014; NCI-2024-04895 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NRG-BN014 (Other: NRG Oncology); NRG-BN014 (Other: CTEP); U10CA180868 (NIH)
Record Dates: First submitted 2024-07-08; First posted 2024-07-15 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Anatomic Stage IV Breast Cancer AJCC v8; Metastatic Breast Carcinoma; Metastatic Lung Non-Small Cell Carcinoma; Metastatic Malignant Neoplasm in the Leptomeninges; Stage IV Lung Cancer AJCC v8
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Non-Small-Cell Lung; Meningeal Carcinomatosis; Lung Neoplasms | interventions — Specimen Handling; Spinal Puncture; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (IFRT) (Active Comparator): Patients undergo involved-field radiation therapy delivered to specific areas of LM that are causing and/or may cause symptoms 5 days a week for a total of 10 days of treatment in the absence of disease progression or unacceptable toxicity. Patients undergo CT or PET/CT during screening and MRI as well as LP throughout the study. Patients may optionally undergo research blood sample and CSF collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Radiation: Involved-Field Radiation Therapy; Procedure: Lumbar Puncture; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Other: Quality-of-Life Assessment
- Arm 2 (pCSI) (Experimental): Patients undergo pCSI radiation therapy delivered to the entire space containing the CSF, brain, and spinal cord 5 days a week for a total of 10 days of treatment in the absence of disease progression or unacceptable toxicity. Patients undergo CT or PET/CT during screening and MRI as well as possible LP throughout the study. Patients may optionally undergo research blood sample and CSF collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Lumbar Puncture; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Radiation: Proton Beam Craniospinal Irradiation; Other: Quality-of-Life Assessment

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood and CSF sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT or PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Radiation: Involved-Field Radiation Therapy — Undergo IFRT
  Other Names: IFRT; Involved field radiotherapy
  Arms: Arm 1 (IFRT)
Procedure: Lumbar Puncture — Undergo LP
  Other Names: LP; Spinal Tap
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Radiation: Proton Beam Craniospinal Irradiation — Undergo pCSI
  Other Names: Craniospinal Proton Beam Radiation Therapy; p-CSI; Proton Craniospinal Irradiation; Proton Craniospinal Radiation Therapy
  Arms: Arm 2 (pCSI)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This phase III trial compares proton craniospinal irradiation (pCSI) to involved-field radiation therapy (IFRT) for the treatment of breast or non-small cell lung cancer that has spread from where it first started to the cerebrospinal fluid filled space that surrounds the brain and spinal cord (leptomeningeal metastasis). Patients with leptomeningeal metastasis (LM) may develop multiple areas of nervous system (neurologic) impairment that can be life-threatening. Radiation therapy (RT) effectively relieves local symptoms due to LM. RT uses high energy radiography (x-rays), particles, or radioactive seeds to kill cancer cells and shrink tumors. IFRT is commonly used to treat symptoms of LM. IFRT is radiation treatment that uses x-rays to treat specific areas of LM and to relieve and/or prevent symptoms. pCSI uses protons that can be directed with more accuracy than x-rays which allows treatment of the entire central nervous system space containing the cerebrospinal fluid (CSF), brain, and spinal cord. The pCSI treatment could delay the worsening of LM. Giving pCSI may be better than IFRT in treating LM in patients with breast or non-small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare overall survival (OS) between proton craniospinal irradiation (pCSI) and involved-field radiotherapy (IFRT) in patients with breast cancer or non-small cell lung cancer (NSCLC) leptomeningeal metastasis.

SECONDARY OBJECTIVES:

I. To compare central nervous system progression-free survival (CNS PFS) between pCSI and IFRT in patients with breast cancer or NSCLC leptomeningeal metastasis.

II. To compare time to CNS progression between pCSI and IFRT in patients with breast cancer or NSCLC leptomeningeal metastasis.

III. To compare CNS PFS between pCSI and IFRT in patients with breast cancer or NSCLC leptomeningeal metastasis, as evaluated by central review of imaging.

IV. To compare the rate of radiation-induced central nervous system necrosis between pCSI versus (vs.) IFRT in patients with breast cancer or NSCLC leptomeningeal metastasis.

V. To characterize treatment-related adverse events using Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0.

VI. To compare patient-reported outcomes (symptoms severity subscale per MD Anderson Symptom Inventory for Brain Tumors [MDASI-BT] and MD Anderson Symptom Inventory for Spine Tumors [MDASI-SP]) in patients with breast cancer or non-small cell lung cancer leptomeningeal metastasis.

EXPLORATORY OBJECTIVE:

I. To compare patient-reported outcomes (symptoms interference, brain tumor-specific, spine tumor-specific subscales per MDASI-BT and MDASI-SP) in patients with breast cancer or non-small cell lung cancer leptomeningeal metastasis.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM 1: Patients undergo involved-field radiation therapy delivered to specific areas of LM that are causing and/or may cause symptoms 5 days a week for a total of 10 days of treatment in the absence of disease progression or unacceptable toxicity. Patients undergo computed tomography (CT) or positron emission tomography (PET)/CT during screening and magnetic resonance imaging (MRI) as well as possible lumbar puncture (LP) throughout the study. Patients may optionally undergo research blood sample and CSF collection throughout the study.

ARM 2: Patients undergo pCSI radiation therapy delivered to the entire space containing the CSF, brain, and spinal cord 5 days a week for a total of 10 days of treatment in the absence of disease progression or unacceptable toxicity. Patients undergo CT or PET/CT during screening and MRI as well as possible LP throughout the study. Patients may optionally undergo research blood sample and CSF collection throughout the study.

After completion of study treatment, patients are followed every 3 months for 12 months, and then every 6 months for up to 3 years from end of RT.

ELIGIBILITY:
Inclusion Criteria:

* PRIOR TO STEP 1 REGISTRATION
* Patients with pathologically (histologically or cytologically) proven diagnosis of breast cancer or NSCLC
* Patients must have newly diagnosed leptomeningeal metastasis established through at least one of the following:

  * Positive CSF cytology for malignancy

    * CSF cytology with suspicious cells is considered positive; CSF cytology with atypical cells is considered equivocal and not positive
  * Patients with an equivocal or negative CSF cytology result, or not suitable for CSF sampling, radiographic diagnosis of leptomeningeal metastasis with linear and/or nodular disease and documentation of typical clinical signs (European Association of Neuro-Oncology [EANO]-European Society for Medical Oncology [ESMO] Diagnostic Criteria Type IIA-IIC) is required

    * Patients with typical clinical signs of leptomeningeal metastasis may have one or more of the following symptoms and signs: headache, nausea, vomiting, mental status change, gait difficulty, cranial nerve palsy, diplopia, visual change, hearing loss, radicular weakness, radicular sensory change, urinary retention, saddle anesthesia, constipation, neck pain, and back pain
  * For patients with prior history of immunotherapy or current immunotherapy, CSF sampling rather than just MRI enhancement is strongly recommended to exclude immune-related aseptic meningitis
* Patients must be candidates for radiation therapy for the treatment of leptomeningeal metastasis
* Age ≥ 18
* PRIOR TO STEP 2 REGISTRATION
* Note: Step 2 registration must occur no later than 30 calendar days after step 1 registration
* Financial clearance for proton therapy treatment
* Patients must have systemic disease evaluation through standard of care imaging for example CT chest/abdomen/pelvis or body PET/CT
* Karnofsky performance status ≥ 60
* Not pregnant and not nursing

  * Negative urine or serum pregnancy test (in persons of childbearing potential) within 14 days prior to registration. Childbearing potential is defined as any person who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) or who is not postmenopausal
* Hemoglobin ≥ 8.0 g/dl (Note: The use of transfusion or other intervention to achieve hemoglobin [Hgb] ≥ 8.0 g/dl is acceptable)
* Absolute neutrophil count (ANC) ≥ 1,000/mm^3 (Note: the use of granulocyte-colony stimulating factor or other intervention to achieve ANC ≥ 1,000/mm^3 is acceptable)
* Platelets ≥ 100,000/mm^3 (Note: the use of transfusion or other intervention to achieve platelets ≥ 100,000/mm^3 is acceptable)
* Total bilirubin ≤ 1.5 × institutional upper limit of normal (ULN) (patients with known Gilbert disease without other clinically significant liver abnormalities are not excluded)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine transaminase (ALT) (serum glutamic pyruvic transaminase [SGPT]) ≤ 3 × ULN
* No prior radiation therapy to the spinal cord with equivalent dose in 2 gray (Gy) fractions (EQD2) more than 40Gy or cauda equina with EQD2 more than 50Gy using alpha/beta ratio of 3
* No prior treatment for leptomeningeal metastasis (note: prior CNS treatment for other non-leptomeningeal disease is allowed)
* No history of unstable angina requiring hospitalization in the last 3 months
* No history of myocardial infarction within the last 3 months
* New York Heart Association Functional Classification II or better (New York Heart Association [NYHA] Functional Classification III/IV are not eligible) (Note: Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification.)
* No active infection currently requiring intravenous (IV) antibiotic management
* No active chronic obstructive pulmonary disease exacerbation or other acute respiratory illness precluding study therapy
* No CTCAE v5.0 ≥ grade 2 encephalopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Estimated)
Dates: Start 2025-03-04 (Actual); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | From randomization until death due to any cause, assessed up to 3 years
  Will be event-driven and will be conducted when a total of 88 OS events (from both treatment arms) have been observed. The final analysis (if the trial does not stop early at an interim) is expected to occur roughly 45 months after study activation (including the initial 6-months ramp-up). All analyses (interim or final) will be done on a modified intent-to-treat (ITT) basis such that all randomized patients who have follow-up information will be included in the arm to which they are randomized regardless of what treatment the patients receive. Treatment comparisons will be based on the log-rank test. At the final analysis, if the test has an associated 1-sided p-value of 0.024 or less in favor of proton craniospinal irradiation (pCSI) (equivalently, Z > 1.98), then the trial will conclude that the pCSI arm results in improved survival over the involved field radiotherapy (IFRT) arm.

SECONDARY OUTCOMES:
Central nervous system (CNS) progression-free survival (PFS) | Randomization until CNS progression or death, whichever occurs first, assessed up to 3 years
  Will be based on modified ITT, including all randomized patients who have follow-up information. The analysis will be performed according to the treatment arm to which patients were randomized. Analysis for CNS-PFS will consist of estimation of its distribution for each treatment arm via the Kaplan-Meier method and a log-rank test. Statistical power will depend on the total CNS-PFS events accumulated at trial end. Additional analyses may consist of estimating the treatment hazard ratio via the Cox proportional hazards model accounting for prognostic covariates including randomization stratification factors evaluating whether the proportional hazards assumption holds or whether any treatment effect is notably time-varying, and evaluating for potential treatment by prognostic covariate interactions.
Time to CNS progression | Randomization until CNS progression, assessed up to 3 years
  Analysis for time to CNS progression will involve comparing the rate of CNS progression in patients who receive pCSI to patients who receive IFRT. The cumulative incidence function (CIF) estimator will be used to estimate the median time to CNS progression in the presence of competing event of deaths in the two arms, separately. The Gray's test will be used to evaluate the difference in the distribution of CNS progression between treatment arms. These results will be interpreted in light of the competing deaths. The comparison of treatment effect on time to CNS progression will involve estimating the cause-specific hazard ratio (CHR) in a Cox proportional hazards model adjusting for patients and disease characteristics (e.g. stratification randomization factors).
Time to radiation-induced CNS necrosis (TTRN) | Randomization until radiation necrosis in brain and/or spinal cord, assessed up to 3 years
  Analysis will involve comparing the rate of radiation necrosis in patients who receive pCSI to patients who receive IFRT. Death will be treated as a competing risk event in this analysis. The cumulative incidence function (CIF) estimator will be used to estimate the median time to radiation-induced CNS necrosis in the presence of competing event of deaths in the two arms, separately. The Gray's test will be used to evaluate the difference in the distribution of TTRN between treatment arms. These results will be interpreted in light of the competing deaths. The comparison of treatment effect on TTRN will involve estimating the CHR in a Cox proportional hazards model adjusting for patients and disease characteristics (e.g. stratification randomization factors).
Incidence of treatment-related adverse events (AEs) | Baseline to 30 days from end of radiation therapy
  Will be evaluated by comparative frequency summaries for all adverse event types between arms. AEs will be graded according to Common Terminology Criteria for Adverse Events version 5.0. Comprehensive summaries of all AEs by treatment arm will be generated and examined. Counts and frequencies of worst (highest score) AE per patient will be presented overall and by AE type category, separately by assigned treatment group. The proportion of patients with at least one grade 3 or higher AE will be compared between treatment arms. Similarly, frequencies for specific potentially treatment related AEs where grade 3 or higher events are noted may be compared. Any frequencies to be tested will be evaluated using the chi-square or exact test as appropriate, with two-sided significance level 0.05.
Patient reported outcomes (PRO) | Baseline to 24 months post-radiation therapy
  Will be assessed using MD Anderson Symptom Inventory for Brain Tumors and MD Anderson Symptom Inventory for Spine Tumors. Data from these four subscales will be analyzed separately. For each subscale, scores from individual questions will be averaged to arrive at a subscale-specific score for each patient. The symptom severity scores, symptom interference scores, and brain tumor-specific and spine tumor-specific scores will be summarized at each assessment timepoint using descriptive statistics and visualized with box plots and series plots. Changes over time will also be assessed visually. The comparison of changes in quality of life between treatment arms will be conducted separately for each of these four subscales using mixed effects models.

OTHER OUTCOMES:
Estimates of the primary outcome treatment effect by sex | Up to 3 years
  Will estimate the primary outcome treatment effect and the corresponding 95% confidence intervals (CIs) by sex.
Estimates of the primary outcome treatment effect by race | Up to 3 years
  Will estimate the primary outcome treatment effect and the corresponding 95% CIs by race.
Estimates of the primary outcome treatment effect by ethnicity | Up to 3 years
  Will estimate the primary outcome treatment effect and the corresponding 95% CIs by ethnicity.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan T Yang, Principal Investigator — NRG Oncology
Locations (57):
- United States (57):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - UC San Diego Health System - Encinitas, Encinitas, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - UC San Diego Medical Center - Hillcrest, San Diego, California
  - California Protons Cancer Therapy Center, San Diego, California
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - UM Sylvester Comprehensive Cancer Center at Aventura, Aventura, Florida
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - UM Sylvester Comprehensive Cancer Center at Doral, Doral, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Miami Cancer Institute, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Kendall, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - Alton Memorial Hospital, Alton, Illinois
  - Northwestern University, Chicago, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Memorial Hospital East, Shiloh, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - McLaren Cancer Institute-Flint, Flint, Michigan
  - Karmanos Cancer Institute at McLaren Greater Lansing, Lansing, Michigan
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - NYU Langone Hospital - Brooklyn, Brooklyn, New York
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - New York Proton Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Inova Alexandria Hospital, Alexandria, Virginia
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - Inova Fair Oaks Hospital, Fairfax, Virginia
  - Inova Loudoun Hospital, Leesburg, Virginia